CLINICAL TRIAL: NCT00706121
Title: S0000D: A Study of the Effect of Vitamin E and/or Selenium on Adenomatous Colorectal Polyps (ACP) in Participants Enrolled in SELECT
Brief Title: S0000D: Effect of Vitamin E and/or Selenium on Colorectal Polyps in Men Enrolled on SELECT Trial SWOG-S0000
Acronym: ACP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000593329; S0000D (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: colon cancer; rectal cancer; adenomatous polyp
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyps | interventions — Vitamin E; alpha-Tocopherol; Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin E + selenium placebo (Experimental): Vitamin E and selenium placebo daily for 7 - 12 years
  Interventions: Drug: Vitamin E; Drug: selenium placebo
- Selenium + vitamin E placebo (Experimental): Selenium and vitamin E placebo daily for 7 - 12 years
  Interventions: Drug: Selenium; Drug: Vitamin E placebo
- Vitamin E + selenium (Experimental): Vitamin E and selenium daily for 7 - 12 years
  Interventions: Drug: Vitamin E; Drug: Selenium
- Vitamin E placebo + selenium placebo (Placebo Comparator): Vitamin E placebo and selenium placebo daily for 7 - 12 years
  Interventions: Drug: Vitamin E placebo; Drug: selenium placebo

INTERVENTIONS:
Drug: Vitamin E — 400 IU daily by mouth for 7 - 12 years
  Other Names: alpha tocopherol
  Arms: Vitamin E + selenium; Vitamin E + selenium placebo
Drug: Selenium — 200 mcg daily for 7 - 12 years
  Other Names: L-selenomethionine
  Arms: Selenium + vitamin E placebo; Vitamin E + selenium
Drug: Vitamin E placebo — 1 pill by mouth daily for 7 - 12 years
  Other Names: placebo
  Arms: Selenium + vitamin E placebo; Vitamin E placebo + selenium placebo
Drug: selenium placebo — 1 pill by mouth daily for 7 - 12 years
  Other Names: placebo
  Arms: Vitamin E + selenium placebo; Vitamin E placebo + selenium placebo

SUMMARY:
RATIONALE: Studying tissue samples in the laboratory from participants receiving treatment on the Selenium and Vitamin E Cancer Prevention Trial (SELECT) SWOG-S0000 may help doctors predict a participant's response to treatment and help plan the best treatment.

PURPOSE: This phase III trial is studying the effect of vitamin E and/or selenium on colorectal polyps in men enrolled on SELECT Trial SWOG-S0000.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of selenium on colorectal adenoma (CRA) occurrence.
* To assess the effect of selenium on number, location, size, histologic type, and degree of dysplasia of CRA.
* To assess the effect of selenium on colorectal cancer (CRC) incidence.

Secondary

* To assess the effect of vitamin E on CRA occurrence.
* To assess the effect of vitamin E on CRC incidence.

Tertiary

* To explore the effect modification of selenium and vitamin E by aspirin on CRA occurrence.
* To explore the effect modification of selenium and vitamin E by body mass index.

OUTLINE: This is a multicenter study.

Endoscopically obtained tissue samples are reviewed by study pathologists to confirm the presence (or absence) of a colorectal adenoma (CRA). If a CRA is present, the number, location, size, histology, and degree of dysplasia are documented. The CRA is also reviewed to exclude a diagnosis of colorectal cancer.

Additional data, including aspirin use, height and weight, date of birth, and other demographic and baseline characteristics, is also obtained. Participants' medical records are reviewed periodically.

Participants are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on the Selenium and Vitamin E Cancer Prevention Trial (SELECT) SWOG-S0000
* Screened by lower endoscopy (i.e., sigmoidoscopy and/or colonoscopy) after randomization on SELECT trial

PATIENT CHARACTERISTICS:

* Willing to sign an applicable medical records release form
* Willing to allow the release of tissue for central pathology review of resected polyps and endoscopic biopsies

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8094 (Actual)
Dates: Start 2008-06; Primary Completion 2015-10 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Peter Lance, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
http://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Derived] Goodman PJ, Tangen CM, Darke AK, Arnold KB, Hartline J, Yee M, Anderson K, Caban-Holt A, Christen WG, Cassano PA, Lance P, Klein EA, Crowley JJ, Minasian LM, Meyskens FL. Opportunities and challenges in incorporating ancillary studies into a cancer prevention randomized clinical trial. Trials. 2016 Aug 12;17:400. doi: 10.1186/s13063-016-1524-9. PMID 27519183

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin E + Selenium Placebo | Selenium + Vitamin E Placebo | Vitamin E + Selenium | Vitamin E Placebo + Selenium Placebo
Started | 2039 | 2096 | 2030 | 1929
Completed | 1643 | 1700 | 1626 | 1577
Not Completed | 396 | 396 | 404 | 352

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E + Selenium Placebo | Selenium + Vitamin E Placebo | Vitamin E + Selenium | Vitamin E Placebo + Selenium Placebo | Total
Number analyzed (Participants) | 1643 | 1700 | 1626 | 1577 | 6546
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.0 [58.0 to 66.0] | 62.0 [58.0 to 66.0] | 62.0 [58.0 to 67.0] | 62.0 [58.0 to 67.0] | 62.0 [58.0 to 66.0]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 50-54 | 60 | 59 | 49 | 52 | 220
  Age, Categorical: 55-64 | 1025 | 1045 | 1002 | 933 | 4005
  Age, Categorical: 65-74 | 494 | 538 | 516 | 524 | 2072
  Age, Categorical: >= 75 | 64 | 58 | 59 | 68 | 249
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 1643 | 1700 | 1626 | 1577 | 6546
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White | 1411 | 1445 | 1412 | 1374 | 5642
  Race/ethnicity: African American | 181 | 187 | 167 | 160 | 695
  Race/ethnicity: Hispanic, not African American | 30 | 30 | 32 | 25 | 117
  Race/ethnicity: Hispanic, African American | 2 | 1 | 1 | 0 | 4
  Race/ethnicity: Aboriginal | 2 | 8 | 1 | 7 | 18
  Race/ethnicity: Asian/Pacific Islander | 12 | 22 | 11 | 9 | 54
  Race/ethnicity: Other | 5 | 7 | 2 | 2 | 16
Education [Count of Participants; unit: Participants] — Population: Subjects missing education information excluded.
  Participants
    <=High school/GED: number analyzed (Participants) | 1639 | 1691 | 1615 | 1572 | 6517
    <=High school/GED | 263 | 264 | 226 | 263 | 1016
    Some college/vocational: number analyzed (Participants) | 1639 | 1691 | 1615 | 1572 | 6517
    Some college/vocational | 432 | 447 | 397 | 378 | 1654
    >=College graduate: number analyzed (Participants) | 1639 | 1691 | 1615 | 1572 | 6517
    >=College graduate | 944 | 980 | 992 | 931 | 3847
Smoking Status [Count of Participants; unit: Participants] — Population: Subjects missing smoking history excluded.
  Participants
    number analyzed (Participants) | 1642 | 1698 | 1625 | 1575 | 6540
    Never | 729 | 785 | 726 | 711 | 2951
    Current | 87 | 98 | 99 | 97 | 381
    Former | 826 | 815 | 800 | 767 | 3208
BMI, Categorical [Count of Participants; unit: Participants] — Population: Subjects missing BMI excluded.
  Participants
    number analyzed (Participants) | 1639 | 1695 | 1619 | 1572 | 6525
    Normal or underweight (<=25) | 293 | 355 | 327 | 324 | 1299
    Overweight (>25 to 30) | 818 | 795 | 800 | 764 | 3177
    Obese (>30) | 528 | 545 | 492 | 484 | 2049
BMI, Continuous [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Subjects missing BMI excluded.
  kg/m^2
    number analyzed (Participants) | 1639 | 1695 | 1619 | 1572 | 6525
    (all) | 27.8 [25.7 to 31.2] | 28.0 [25.4 to 30.9] | 27.8 [25.6 to 30.9] | 28.0 [25.4 to 30.8] | 27.9 [25.7 to 30.9]
History of Cancer [Count of Participants; unit: Participants] | 38 | 32 | 35 | 30 | 135
History of Colorectal Cancer [Count of Participants; unit: Participants] | 7 | 7 | 7 | 5 | 26
History of Colon Polyps [Count of Participants; unit: Participants] | 355 | 347 | 339 | 355 | 1396
History of Diverticulitis [Count of Participants; unit: Participants] | 128 | 103 | 121 | 110 | 462
History of Diabetes [Count of Participants; unit: Participants] | 138 | 126 | 126 | 148 | 538
Number of First Degree Relatives with Colorectal Cancer [Count of Participants; unit: Participants] — Population: Subjects missing FDR information excluded.
  Participants
    number analyzed (Participants) | 1560 | 1617 | 1554 | 1501 | 6232
    0 | 1347 | 1393 | 1350 | 1279 | 5369
    1 | 185 | 198 | 181 | 196 | 760
    2 or more | 28 | 26 | 23 | 26 | 103
Medication Use -- Aspirin [Count of Participants; unit: Participants] | 756 | 769 | 775 | 736 | 3036
Medication Use -- Cox II Inhibitors [Count of Participants; unit: Participants] — Population: Subjects missing information on Cox II inhibitor use excluded.
  Participants
    number analyzed (Participants) | 1641 | 1697 | 1624 | 1575 | 6537
    (all) | 91 | 85 | 92 | 77 | 345
Medication Use -- Other NSAIDs [Count of Participants; unit: Participants] — Population: Subjects missing information on NSAID use excluded.
  Participants
    number analyzed (Participants) | 1641 | 1698 | 1626 | 1576 | 6541
    (all) | 173 | 175 | 164 | 168 | 680
Medication Use -- Statins [Count of Participants; unit: Participants] — Population: Subjects missing information on or not asked about statin use excluded.
  Participants
    number analyzed (Participants) | 992 | 1050 | 1005 | 955 | 4002
    (all) | 280 | 297 | 283 | 284 | 1144

OUTCOME MEASURES:

1. Primary Outcome: Effect of Selenium on Colorectal Adenoma (CRA) Occurrence, Analyzed by Active Selenium vs. Selenium Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo selenium.
Measure: Count of Participants; unit: Participants
Groups:
- Active Selenium: Active Selenium +/- Vitamin E
- Selenium Placebo: Selenium Placebo +/- Vitamin E
Arm/Group | Active Selenium | Selenium Placebo
Number analyzed (Participants) | 3326 | 3220
Participants | 1136 | 1150
Statistical Analysis 1: Comparison: Active Selenium vs Selenium Placebo; Test type: Superiority or Other; p = 0.96, Log binomial regression; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.9 to 1.02]

2. Primary Outcome: Effect of Selenium on Advanced Neoplasia, Analyzed by Active Selenium vs. Selenium Placebo
Description: Adenomas with diameter >=1cm or any adenoma with villous features or high-grade dysplasia
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo selenium.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Selenium | Selenium Placebo
Number analyzed (Participants) | 3326 | 3220
Participants | 269 | 282
Statistical Analysis 1: Comparison: Active Selenium vs Selenium Placebo; Test type: Superiority or Other; p = 0.32, Log binomial regression; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.78 to 1.08]

3. Primary Outcome: Effect of Selenium and/or Vitamin E on Colorectal Cancer (CRC) Incidence
Time Frame: From 1 year post randomization through study completion
Measure: Count of Participants; unit: Participants
Groups:
- Vitamin E: Vitamin E + matching placebo for selenium
- Selenium: Selenium + matching placebo for vitamin E
- Combination: Vitamin E + selenium
- Placebo: Matching placebo for vitamin E + matching placebo for selenium
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 1643 | 1700 | 1626 | 1577
Participants | 10 | 11 | 9 | 6

4. Primary Outcome: Effect of Selenium on Occurrences of Multiple (>2) Adenomas
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo selenium.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Selenium | Selenium Placebo
Number analyzed (Participants) | 3326 | 3220
Participants | 258 | 276
Statistical Analysis 1: Comparison: Active Selenium vs Selenium Placebo; Test type: Superiority or Other; p = 0.24, Log binomial regression; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.77 to 1.07]

5. Secondary Outcome: Effect of Vitamin E on CRA Occurrence, Analyzed by Active Vitamin E vs. Vitamin E Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo Vitamin E.
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin E: Active vitamin E +/- selenium
- Vitamin E Placebo: Vitamin E placebo +/- selenium
Arm/Group | Active Vitamin E | Vitamin E Placebo
Number analyzed (Participants) | 3269 | 3277
Participants | 1159 | 1127
Statistical Analysis 1: Comparison: Active Vitamin E vs Vitamin E Placebo; Test type: Superiority or Other; p = 0.38, Log binomial regression; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.96 to 1.10]

6. Other Pre Specified Outcome: Effect Modification of Selenium by Body Mass Index on CRA Occurrence, Analyzed by Active Selenium vs. Selenium Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo selenium.
Measure: Number; unit: percentage of participants
Arm/Group | Active Selenium | Selenium Placebo
Number analyzed (Participants) | 1133 | 1146
percentage of participants
  Normal | 30.2 | 31.4
  Overweight | 35.2 | 36.5
  Obese | 35.2 | 37.0

7. Other Pre Specified Outcome: Effect Modification of Selenium by Aspirin on CRA Occurrence, Analyzed by Active Selenium vs. Selenium Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo selenium.
Measure: Number; unit: ercentage of participants in subgroup
Arm/Group | Active Selenium | Selenium Placebo
Number analyzed (Participants) | 1136 | 1150
ercentage of participants in subgroup
  Users | 33.5 | 36.4
  Non-users | 34.9 | 34.9

8. Other Pre Specified Outcome: Effect Modification of Vitamin E by Body Mass Index on CRA Occurence, Analyzed by Active Vitamin e vs. Vitamin e Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo Vitamin E.
Measure: Number; unit: ercentage of participants in subgroup
Arm/Group | Active Vitamin E | Vitamin E Placebo
Number analyzed (Participants) | 1155 | 1124
ercentage of participants in subgroup
  Normal | 30.2 | 31.4
  Overweight | 36.8 | 34.9
  Obese | 36.5 | 35.7

9. Other Pre Specified Outcome: Effect Modification of Vitamin E by Aspirin on CRA Occurrence, Analyzed by Active Vitamin e vs. Vitamin e Placebo
Time Frame: From 1 year post randomization through study completion
Population: Marginal analyses were performed, with arms pooled based on active vs. placebo Vitamin E.
Measure: Number; unit: ercentage of participants in subgroup
Arm/Group | Active Vitamin E | Vitamin E Placebo
Number analyzed (Participants) | 1159 | 1127
ercentage of participants in subgroup
  Users | 34.5 | 35.3
  Non-users | 36.5 | 33.3

ADVERSE EVENTS:
Time Frame: Every 6 months while the participant is receiving study supplements.
Description: There are no Adverse Events (AE) associated with this trial. All AEs were reported for the parent trial (SELECT - S0000). Included below are the AEs for the participants on this trial that were included in the primary analysis. These AEs were also reported for the parent trial.
Arm/Group | Vitamin E + Selenium Placebo | Selenium + Vitamin E Placebo | Vitamin E + Selenium | Vitamin E Placebo + Selenium Placebo
Serious Adverse Events (participants affected / at risk) | 10/1643 | 12/1700 | 14/1626 | 19/1577
Other Adverse Events (participants affected / at risk) | 116/1643 | 85/1700 | 112/1626 | 100/1577
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin E + Selenium Placebo (N=1643) | Selenium + Vitamin E Placebo (N=1700) | Vitamin E + Selenium (N=1626) | Vitamin E Placebo + Selenium Placebo (N=1577)
Cardiac ischemia/infarction (Cardiac disorders) | 2 | 5 | 7 | 6
Cardiovascular-other (Cardiac disorders) | 3 | 3 | 6 | 6
Supraventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Surgery-hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 0 | 1
CNS hemorrhage (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebrovascular ischemia (Nervous system disorders) | 2 | 2 | 3 | 2
Erectile impotence (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Carotid stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial ischemia (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin E + Selenium Placebo (N=1643) | Selenium + Vitamin E Placebo (N=1700) | Vitamin E + Selenium (N=1626) | Vitamin E Placebo + Selenium Placebo (N=1577)
Cardiac ischemia/infarction (Cardiac disorders) | 116 | 85 | 112 | 100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less